CLINICAL TRIAL: NCT00037128
Title: Study of GL701 in Men With Systemic Lupus Erythematosus
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Genelabs Technologies (Industry)
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: GL97-01
Record Dates: First submitted 2002-05-16; First posted 2002-05-17 (Estimated); Last update posted 2005-06-24 (Estimated); Status verified 2004-05

CONDITIONS: Systemic Lupus Erythematosus
Keywords: Lupus; SLE; DHEA; GL701
MeSH Terms: conditions — Lupus Erythematosus, Systemic

INTERVENTIONS:
Drug: GL701

SUMMARY:
Lupus flares and other symptoms associated with systemic lupus erythematosus (SLE) may be caused by a deficiency of dehydroepiandrosterone (DHEA). GL701 is an investigational new drug meant to enhance DHEA levels. This study is designed to evaluate both the safety and efficacy of GL701 in male lupus patients.

ELIGIBILITY:
Inclusion Criteria

* Patient must have a diagnosis of SLE > 6 months according to the 1989 revised ACR criteria. Patient must meet at least four of the eleven ACR criteria for systemic lupus
* Patient must have a modified SLEDAI score > 3 at both screening and qualifying visits (Appendix A-2)
* Patient must be treated for SLE with doses of prednisone < 30 mg/day (including those on NO glucocorticoid therapy) unchanged for > 6 weeks prior to study entry (including both screening and qualifying visits). Prednisone dose in patient's receiving alternate day therapy will be the mean daily prednisone dose
* Patient treated with azathioprine, methotrexate, or hydrochloroquine must be on a stable dose with no change in dose for at least 6 weeks preceding the study
* Patient must be able to read and speak English and willing to sign an informed consent in English

Exclusion Criteria

* Patient with a history of prostate cancer
* Patient with elevated Prostate Specific Antigen (PSA)
* Patient diagnosed with liver disease, defined as AST or ALT > 3x the upper limit of normal
* Patient ingesting body building/anabolic steroids within the last 6 months preceding the study
* Patient with end stage renal disease or receiving hemodialysis treatment
* Patient with serum creatinine > 2 mg/dl or creatinine clearance < 60 ml/min
* Patient receiving treatment with ACTH within the 3 months preceding study entry
* Patient receiving androgens, immunoglobulins, cyclophosphamide, cyclosporin A, or other immunosuppressive agents, except azathioprine, methotrexate, and hydrochloroquine within the last 3 months
* Patient with known hypersensitivity to DHEA or the inactive ingredients used in the GL70l formulation (cornstarch, lactose, and magnesium stearate)
* Patient who participated in any prior DHEA study or administration of DHEA within the past 3 months
* Patient using any investigational agents within the longer of 30 days or 10 half-lives of the agent
* Patient with any condition which in the Investigator's or sponsor's opinion is sufficient to prevent adequate compliance with the study or likely to confuse follow-up evaluation (e.g.. alcoholism, drug addiction, acute withdrawal from chemical dependency, psychiatric disease)
* Patient requires treatment/medication prohibited by protocol
* Patient with any serious EKG abnormality as determined by the Investigator

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40
Dates: Start 1998-03

CONTACTS AND LOCATIONS:
Locations (1):
- Genelabs Technologies, Inc., Redwood City, California, United States